CLINICAL TRIAL: NCT04291742
Title: Prospective and Randomized Study to Compare the Efficacy of Cognitive Fusion Prostate Biopsies and Prostate Biopsies Performed by "BK-fusion®" Software, for the Diagnosis of Significant Prostate Cancer
Brief Title: Comparison of Prostate Fusion Biopsies With Software and Cognitive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)161/2019
Record Dates: First submitted 2020-02-02; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer Detection; Fusion Prostate Biopsy
Keywords: prostate biopsy; mpMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0: cognitive (Experimental): target prostate biopsies by cognitive fusion
  Interventions: Diagnostic Test: cognitive vs software
- 1: software (Experimental): target prostate biopsies by software
  Interventions: Diagnostic Test: cognitive vs software

INTERVENTIONS:
Diagnostic Test: cognitive vs software — cognitive vs software

SUMMARY:
This study evaluates the efficacy to diagnose significant prostate cancer in patients with suspicious lesions in mpMRI (multiparametric magnetic resonance imaging) by comparing prostate biopsies performed by cognitive fusion with respect to those performed with software fusion (BK-fusion®). Half of the patients included will undergo a systematic prostate biopsy + target biopsies by cognitive fusion and the other half of the population, will undergo a systematic prostate biopsy + target biopsies by software fusion.

DETAILED DESCRIPTION:
Various techniques have been developed to perform targeted prostate biopsies aimed at suspicious lesions detected in mpMRI. The two most frequently used are cognitive fusion, in which the physician locates the areas where the mpMRI detects suspicious lesions and directs the puncture by ultrasound; and software fusion, in which the images of the mpMRI are integrated by a software with the ultrasound allowing to direct the puncture to the lesion itself. Both forms of fusion biopsy have proven to be superior to systematized prostate biopsies in the detection of significant prostate cancer, although neither has demonstrated superiority over the other.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years.
* mpMRI carried out in our center.
* Presence of lesions with PIRADSv.2 ≥ 3.
* Acceptance to participate in the study.

Exclusion Criteria:

* PSA> 30 ng / ml
* Treatment with 5-ARIs (5-alpha-reductase inhibitors).
* Previous diagnosis of PCa.
* TR> T3.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-02-27 (Estimated); Study Completion 2022-02-27 (Estimated)

PRIMARY OUTCOMES:
Rate of overall prostate cancer and significant prostate cancer between the groups | 2 years
  Differences in percentage of detection of overall prostate cancer and prostate cancer ISUP equal or greater than 2 between both groups will be assessed.

SECONDARY OUTCOMES:
Rate of overall prostate cancer and significant prostate cancer between the groups according to the location of the lesions. | 2 years
  Differences in percentage of detection of overall prostate cancer and prostate cancer ISUP equal or greater than 2 between both groups will be assessed according to the location of the lesions.
Rate of overall prostate cancer and significant prostate cancer between the groups according to the size of the lesions. | 2 years
  Differences in percentage of detection of overall prostate cancer and prostate cancer ISUP equal or greater than 2 between both groups will be assessed according to the size of the lesions.
Rate of overall prostate cancer and significant prostate cancer between the groups according to the PIRADS (prostate imaging and reporting and data System) of the lesions. | 2 years
  Differences in percentage of detection of overall prostate cancer and prostate cancer ISUP equal or greater than 2 between both groups will be assessed according to the PIRADS (prostate imaging and reporting and data System) of the lesions.
Rate of overall prostate cancer and significant prostate cancer between the groups according to the prostate volume. | 2 years
  Differences in percentage of detection of overall prostate cancer and prostate cancer ISUP equal or greater than 2 between both groups will be assessed according to the prostate volume.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Celma, MD, Principal Investigator — Hospital Vall d'Hebron, Barcelona
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No